CLINICAL TRIAL: NCT02416310
Title: Effect of Perioperative Transcutaneous Electrical Acupoint Stimulation on Gastrointestinal Function After Cesarean Section
Brief Title: Transcutaneous Electrical Acupoint Stimulation on Gastrointestinal Function After Cesarean Section
Acronym: TEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Principal Investigator, wangqiang, professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Xijing H; mazuike (Other: Xijing Hospital)
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Cesarean Section
Keywords: TEAS; cesarean section; gastrointestinal function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TEAS group (Experimental): TEAS are performed by a specific investigator on the specially acupoint.
  Interventions: Device: TEAS
- Sham group (Sham Comparator): TEAS are performed by a specific investigator on the non-acupoint.
  Interventions: Device: TEAS
- Control group (Placebo Comparator): Only place cutted electrodes but do not give any electrical stimulation.
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — According to ancient Chinese medical books, acupoints SP6 and ST36 are chosen and identified.The patients in TEAS group received electrical stimulation with the 'disperse-dense' waves. Non-acupoint is located 2cm interior to the ST36 and SP6.For group TEAS and Sham, TEAS will be administered 30 minutes prior to surgery and continued until the end of the surgery.Control patients will receive the same treatment without electrical stimulation.
  Other Names: Transcutaneous electrical acupoint stimulation

SUMMARY:
To determine whether treating by transcutaneous electrical acupoint stimulation (TEAS) during perioperative could alleviate the postoperative gastrointestinal complications after cesarean section under combined spinal epidural anesthesia compared with control and non-acupoint group.

DETAILED DESCRIPTION:
Acupuncture is a traditional Chinese medical technique that involves the insertion of needles at acupoints to treat diseases.Clinical evidence supports the efficacy of acupuncture treatment in many applications. Some previous studies reported that stimulation at some acupoint exerted good effects on the digestive system.Compared with acupuncture, transcutaneous electric acupoint stimulation(TEAS) is a non-invasive technique that has similar effects to acupuncture.We hypothesize that TEAS before anesthesia and during surgery would decrease the morbidity and mortality of postoperative complications in 30 days after Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status 1or2, scheduled for elective cesarean section under combined spinal epidural anesthesia
2. Gestational age ≥38 weeks
3. Provide written informed consent

Exclusion Criteria:

1. ASA status≥Ⅲ
2. Patients undergoing surgery within 12 h of admission to hospital
3. Patients with fetal anomaly，medical or obstetric complications such as Diabetes mellitus、Hypertension、Obesity(BMW≥35)
4. Patients suffered from drug addiction or impaired mental state
5. Patients who have a history of gastrointestinal surgery or chronic gastrointestinal disease.
6. Patients with contraindications to the use of electro-acupuncture, such as skin damage or infection at the acupoints
7. Patients with experience of transcutaneous electrical stimulation treatment
8. Participate in the other clinical trial 3 months before the enrollment
9. Not suitable to participate in this experiment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-26 (Actual)

PRIMARY OUTCOMES:
Time to the presence of bowel sound, time to the first passage of flatus, time to the first passage of stool , time to the start of regular diet | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  This is a composite outcome to estimate the gastrointestinal motility function

SECONDARY OUTCOMES:
Electrogastrogram | The first and second days after surgery
Rate of nausea, vomiting, cramping abdominal pain, abdominal distension | Participants will be followed for the duration of hospital stay, an expected average of 5 days
  This is a composite outcome to estimate the complication of digestive system
length of postoperative hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 5 days
Quality of life during 30 days after surgery | One month
  This is a scale to evaluate the quality of life after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Study Chair — Xijing Hospital

REFERENCES:
- [Background] Larson JD, Gutowski KA, Marcus BC, Rao VK, Avery PG, Stacey DH, Yang RZ. The effect of electroacustimulation on postoperative nausea, vomiting, and pain in outpatient plastic surgery patients: a prospective, randomized, blinded, clinical trial. Plast Reconstr Surg. 2010 Mar;125(3):989-94. doi: 10.1097/PRS.0b013e3181ccdc23. PMID 20195124
- [Background] Kotani N, Hashimoto H, Sato Y, Sessler DI, Yoshioka H, Kitayama M, Yasuda T, Matsuki A. Preoperative intradermal acupuncture reduces postoperative pain, nausea and vomiting, analgesic requirement, and sympathoadrenal responses. Anesthesiology. 2001 Aug;95(2):349-56. doi: 10.1097/00000542-200108000-00015. PMID 11506105
- [Background] Cheong KB, Zhang JP, Huang Y. The effectiveness of acupuncture in postoperative gastroparesis syndrome--a systematic review and meta-analysis. Complement Ther Med. 2014 Aug;22(4):767-86. doi: 10.1016/j.ctim.2014.05.002. Epub 2014 May 12. PMID 25146082
- [Background] Oshima M, Aoyama K, Warabi K, Akazawa T, Inada E. Electrogastrography during and after cesarean delivery. J Anesth. 2009;23(1):75-9. doi: 10.1007/s00540-008-0692-5. Epub 2009 Feb 22. PMID 19234827
- [Background] Dresang LT, Leeman L. Cesarean delivery. Prim Care. 2012 Mar;39(1):145-65. doi: 10.1016/j.pop.2011.11.007. PMID 22309587